CLINICAL TRIAL: NCT00175929
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, 3 Parallel Groups, Dose-ranging Trial Evaluating the Efficacy and Safety of Ucb 34714 Used as Adjunctive Treatment at Doses of 50 and 150 mg/Day in b.i.d. Administration (Oral Capsules of 25 mg) for a Maximum of 12 Weeks in Subjects From 16 to 65 Years With Refractory Epilepsy Suffering From Partial Onset Seizures Whether or Not Secondarily Generalized
Brief Title: A Study of Brivaracetam in Subjects With Partial Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01114; 2004-001856-35 (EudraCT Number)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Epilepsy, Focal
Keywords: Epilepsy; Focal Epilepsy; Partial Onset Seizures; Brivaracetam
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo tablets administered twice a day
  Interventions: Other: Placebo
- Brivaracetam 50 mg/day (Experimental): Brivaracetam 50 mg/day, 25 mg administered twice a day
  Interventions: Drug: Brivaracetam
- Brivaracetam 150 mg/day (Experimental): Brivaracetam 150 mg/day, 75 mg administered twice a day
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Other: Placebo — Daily oral dose of two equal intakes, morning and evening, of placebo in a double-blinded way for the 10-week Treatment Period (3 weeks up-titration followed by 7-week maintenance period)
  Arms: Placebo
Drug: Brivaracetam — Daily oral dose of two equal intakes, morning and evening, of Brivaracetam 50 mg/day in a double-blinded way for the 10-week Treatment Period (3 weeks up-titration followed by 7-week maintenance period)
  Arms: Brivaracetam 50 mg/day
Drug: Brivaracetam — Daily oral dose of two equal intakes, morning and evening, of Brivaracetam 150 mg/day in a double-blinded way for the 10-week Treatment Period (3 weeks up-titration followed by 7-week maintenance period)
  Arms: Brivaracetam 150 mg/day

SUMMARY:
This trial will evaluate the efficacy and safety of brivaracetam (at doses of 50 and 150 mg/day in twice a day administration) as add on therapy in subjects with focal epilepsy

ELIGIBILITY:
Inclusion Criteria:

* Well-characterized focal epilepsy or epileptic syndrome according to the International League Against Epilepsy (ILAE) classification
* Subjects with a history of partial onset seizures
* Subjects having at least 4 partial onset seizures during the Baseline period and at least 2 partial onset seizures per month during the 3 months preceding Visit 1
* Subjects being uncontrolled while treated by 1 or 2 concomitant Antiepileptic drug(s) AED(s) being stable
* Male/ female subjects from 16 to 65 years, both inclusive. Subjects under 18 years may only be included where legally permitted and ethically accepted

Exclusion Criteria:

* Seizure type IA non-motor as only seizure type
* History or presence of seizures occurring only in clustered patterns
* History of cerebrovascular accident (CVA)
* Presence of any sign suggesting rapidly progressing brain disorder or brain tumor

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2005-05; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Partial onset seizure frequency (Type I) per week over the 7-week maintenance period | 7-week maintenance period
  Partial onset seizure frequency (Type I) per week over the 7-week maintenance period

SECONDARY OUTCOMES:
Seizure frequency per week for all seizures (types I+II+III) over the 7-week Maintenance period | During the Maintenance period (approximately 7 weeks)
Percentage of reduction from Baseline in seizure frequency per week for partial onset seizures (type I) over the 7-week Maintenance period | During the Maintenance period (approximately 7 weeks)
Percentage of reduction from Baseline in seizure frequency per week for all seizures (types I+II+III) over the 7-week Maintenance period | During the Maintenance period (approximately 7 weeks)
Responder rate in partial onset seizures (type I) over the 7-week Maintenance period | During the Maintenance period (approximately 7 weeks)
  A responder was defined as a subject with a ≥ 50% reduction in seizure frequency per week from the Baseline period to the Maintenance period.
Response to treatment in partial onset seizures (type I) over the 7-week Maintenance period | During the Maintenance period (approximately 7 weeks)
  The percentage reduction from Baseline in partial seizure frequency per week over the Maintenance period was grouped in 5 categories: < -25%, -25% to < 25%, 25% to < 75%, 75% to ≤ 100%, and 100%.
Percentage of seizure-free subjects over the 7-week Maintenance period | During the Maintenance period (approximately 7 weeks)
Percentage of seizure-free days per 4 weeks over Baseline and Maintenance periods | Baseline through Maintenance period (approximately 11 weeks)
Time to N-th seizure in the Maintenance period | During the Maintenance period (approximately 7 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (56):
- Belgium (6):
  - Bruges
  - Brussels
  - Duffel
  - Edegem
  - Leuven
  - Liège
- Czechia (4):
  - Beroun
  - Brno
  - České Budějovice
  - Prague
- Finland (3):
  - Kuopio
  - Oys (Oulu)
  - Tampere
- France (14):
  - Angers
  - Béthune
  - Dijon
  - Grenoble
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Nancy
  - Paris
  - Rennes
  - Strasbourg
  - Tain-l'Hermitage
  - Toulouse
- Germany (11):
  - Berlin
  - Bielefeld
  - Bonn
  - Chemnitz
  - Erlangen
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Kehl
  - München
  - Ulm
- Netherlands (2):
  - Heemstede
  - Heeze
- Poland (6):
  - Gdansk
  - Katowice
  - Lodz
  - Lublin
  - Szczecin
  - Warsaw
- Spain (3):
  - Madrid
  - Valencia
  - Vigo
- United Kingdom (7):
  - Bucks
  - Cambridge
  - Cardiff
  - Glasgow
  - Hartshill
  - Liverpool
  - Newcastle

REFERENCES:
- [Derived] Bresnahan R, Panebianco M, Marson AG. Brivaracetam add-on therapy for drug-resistant epilepsy. Cochrane Database Syst Rev. 2022 Mar 14;3(3):CD011501. doi: 10.1002/14651858.CD011501.pub3. PMID 35285519
- [Derived] Ben-Menachem E, Baulac M, Hong SB, Cleveland JM, Reichel C, Schulz AL, Wagener G, Brandt C. Safety, tolerability, and efficacy of brivaracetam as adjunctive therapy in patients with focal seizures, generalized onset seizures, or Unverricht-Lundborg disease: An open-label, long-term follow-up trial. Epilepsy Res. 2021 Feb;170:106526. doi: 10.1016/j.eplepsyres.2020.106526. Epub 2020 Dec 4. PMID 33461041
- [Derived] Brandt C, Klein P, Badalamenti V, Gasalla T, Whitesides J. Safety and tolerability of adjunctive brivaracetam in epilepsy: In-depth pooled analysis. Epilepsy Behav. 2020 Feb;103(Pt A):106864. doi: 10.1016/j.yebeh.2019.106864. Epub 2020 Jan 12. PMID 31937513
- [Derived] Van Paesschen W, Hirsch E, Johnson M, Falter U, von Rosenstiel P. Efficacy and tolerability of adjunctive brivaracetam in adults with uncontrolled partial-onset seizures: a phase IIb, randomized, controlled trial. Epilepsia. 2013 Jan;54(1):89-97. doi: 10.1111/j.1528-1167.2012.03598.x. Epub 2012 Jul 19. PMID 22813235